CLINICAL TRIAL: NCT04457427
Title: Prospective, Single-center, Randomized Clinical Study to Investigate the Safety and Performance of Diaphragm Stimulation Coupled With Mechanical Ventilation
Brief Title: Randomized Study to Investigate the Safety and Performance of Diaphragm Stimulation Coupled With Mechanical Ventilation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not started
Sponsor: Synapse Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CLIN 20-1000-35
Record Dates: First submitted 2020-03-26; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-03

CONDITIONS: Diaphragm Issues; Ventilator-Induced Lung Injury; Tracheostomy
Keywords: Mechanical Ventilators; Ventilators, Pulmonary; Failure to wean; Lung Injury, Ventilator-Induced; Tracheostomy; Diaphragm pacing
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tracheostomy, no DPS (No Intervention): 5 patients undergoing tracheostomy for failure to wean will receive no additional intervention.
- Trachesotomy with immediate DPS stimulation and monitoring (Experimental): 5 patients undergoing tracheostomy for failure to wean will have DPS implanted concurrently and receive immediate stimulation and monitoring.
  Interventions: Device: NeuRx Diaphragm Pacing System (DPS)
- Trachesotomy with DPS monitoring, stimulation on day 5 (Active Comparator): 5 patients undergoing tracheostomy for failure to wean will have DPS implanted concurrently and receive immediate monitoring followed by stimulation on day 5 post-procedure.
  Interventions: Device: NeuRx Diaphragm Pacing System (DPS)

INTERVENTIONS:
Device: NeuRx Diaphragm Pacing System (DPS) — 4 electrodes are implanted into the diaphragm, 2 on each side, during the tracheostomy procedure. The electrodes are connected to the NeuRx external stimulator which will be used to stimulate and monitor diaphragm activity.
  Arms: Trachesotomy with DPS monitoring, stimulation on day 5; Trachesotomy with immediate DPS stimulation and monitoring

SUMMARY:
This study is a randomized prospective, single-center feasibility study of the use and benefits of NeuRx DPS in patients undergoing tracheostomy for failure to wean.

DETAILED DESCRIPTION:
15 patients undergoing tracheostomy for failure to wean will be randomized into one of 3 cohorts (5 in each cohort): Cohort A: tracheostomy with no intervention; Cohort B: tracheostomy with DPS implantation and immediate stimulation and monitoring and Cohort C: tracheostomy with DPS implantation with monitoring followed with stimulation on day 5.

ELIGIBILITY:
Inclusion Criteria:

* Patient is intubated, on mechanical ventilation, undergoing tracheostomy, and expected to undergo mechanical ventilation for at least 5 days
* Signed written informed consent has been obtained prior to performing any study related procedure(s)
* Subject is at least 18 years of age
* Negative pregnancy test if the patient is a female of child-bearing potential. (Females of child-bearing potential exclude women who are post-hysterectomy or post-menopausal.)

Exclusion Criteria:

* Diaphragm malformation which makes electrode insertion impossible
* Presence of an implantable cardioverter-defibrillator
* Severe chronic obstructive pulmonary disease (COPD)
* Subject is pregnant or breastfeeding
* Diagnosis of neuromuscular disease or high level spinal cord injury prior to tracheostomy
* Terminal patients expected to die during their stay in the hospital
* Participation in other clinical studies that could interfere with the results in the ongoing study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Device and procedure safety | Through study completion, an average of 6 years
  Device or procedure-related adverse events from time of implant until removal of electrodes prior to discharge from the hospital or 30 days, whichever occurs first
Monitoring | Through study completion, an average of 6 years
  Detection of rhythmic diaphragm burst activity for identifying the level of diaphragm dysfunction
Stimulation | Through study completion, an average of 6 years
  Increase in magnitude of diaphragm burst activity with stimulation

SECONDARY OUTCOMES:
Effects of diaphragm stimulation | Through study completion, an average of 6 years
  Effects of diaphragm stimulation on ventilator parameters (plateau pressure, compliance, tidal volumes), oxygenation, weaning time, extubation failure, and length of stay

OTHER OUTCOMES:
Electrode removal | Through study completion, an average of 6 years
  (3) Safe and complete removal of electrodes prior to discharge from the hospital or thirty (30) days, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Tunç Laçin, MD, Principal Investigator — Marmara University
Locations (1):
- Marmara Univeristy, Istanbul, Turkey (Türkiye)

REFERENCES:
- See also: Click here for more information about the Sponsor. — http://www.synapsebiomedical.com/